CLINICAL TRIAL: NCT06622564
Title: Decreasing Postoperative Blood Loss and Seizures by Timing of Intravenous Tranexamic Acid in Open Cardiac Surgery (DEPOSITION)-2 Pilot Trial
Brief Title: Decreasing Postoperative Blood Loss and Seizures by Timing of Intravenous Tranexamic Acid 2 Pilot Trial
Acronym: DEPOSITION-2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEPOSITION-2_2024
Record Dates: First submitted 2024-09-25; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Bleeding; Surgical Blood Loss; Seizures
Keywords: cardiac surgery; tranexamic acid; cardiopulmonary bypass; seizure; blood transfusion
MeSH Terms: conditions — Hemorrhage; Blood Loss, Surgical; Seizures | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: After CPB Tranexamic Acid + Before CPB Placebo versus Before CPB Tranexamic Acid + After CPB Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- After CPB Tranexamic Acid/Placebo (Active Comparator): In the intervention group, patients will receive intravenous administration (10-100 mL of saline placebo) at the induction of anesthesia as a bolus and/or continuous infusion. In addition, patients will receive intravenous administration (5 g of TxA) after heparin reversal (i.e., after CPB).
  Interventions: Drug: After CPB Tranexamic Acid; Drug: Before CPB Placebo
- Before CPB Tranexamic Acid/Placebo (Active Comparator): In the control group, patients will receive an intravenous administration (1-10 g of TxA) at the induction of anesthesia as a bolus and/or continuous infusion (i.e., before CPB). In addition, patients will receive an intravenous administration (50 mL of saline placebo) after heparin reversal.
  Interventions: Drug: Before CPB Tranexamic Acid; Drug: After CPB Placebo

INTERVENTIONS:
Drug: Before CPB Tranexamic Acid — Tranexamic acid 1 to 10 g (10 to 100 mL) administered intravenously as per standard care at the induction of anesthesia as a bolus and/or continuous infusion (i.e., before CPB).
  Other Names: Cyklokapron
  Arms: Before CPB Tranexamic Acid/Placebo
Drug: After CPB Tranexamic Acid — Tranexamic acid 5 g (50 mL) administered after heparin reversal (i.e., after CPB).
  Other Names: Cyklokapron
  Arms: After CPB Tranexamic Acid/Placebo
Drug: Before CPB Placebo — Placebo (10 to 100 mL saline) administered intravenously at the induction of anesthesia as a bolus and/or continuous infusion.
  Other Names: Saline
  Arms: After CPB Tranexamic Acid/Placebo
Drug: After CPB Placebo — Placebo (50 mL saline) administered after heparin reversal.
  Other Names: Saline
  Arms: Before CPB Tranexamic Acid/Placebo

SUMMARY:
The goal of this clinical trial is to establish the feasibility of conducting a large trial to determine the optimal timing of intravenous tranexamic acid administration in cardiac surgery. The main questions it aims to answer are:

* Is it feasible to conduct a larger definitive trial?
* Can we measure the systemic tranexamic acid concentration and fibrinolytic potential in the blood samples?

Researchers will compare intravenous tranexamic acid administered before cardiopulmonary bypass versus after cardiopulmonary bypass to see if the systemic tranexamic acid concentration and fibrinolytic potential are similar or better.

Participants will:

* Provide written informed consent
* Receive tranexamic acid during surgery
* Provide blood samples at 5 time points: before surgery, on arrival in intensive care unit, 3 hours after arrival, 6 hours after arrival, and on the next morning.

DETAILED DESCRIPTION:
Postoperative bleeding related to open cardiac surgery increases the rates of complications and mortality. It results from the blood thinners that are needed for use. Intravenous tranexamic acid (TxA) has become a mainstay in cardiac surgical procedures for decreasing bleeding and minimizing transfusion requirements. Although intravenous TxA is usually well tolerated, there is a well-known risk (1 to 4%) of postoperative seizures. This is due to the similarity between TxA and the brain tissues. The aim is to eliminate the risk of seizures and to improve the protection against bleeding. When TxA is used before and during cardiopulmonary bypass (CPB), the presence of systemic TxA during de-airing of the heart and the termination of CPB may facilitate entry of TxA into the brain causing seizures. Administration of TxA after CPB may result in higher systemic concentrations that may be more effective for protecting against bleeding after surgery. The aim is to establish the feasibility of a definitive trial to prove that administration of TxA after CPB can eliminate postoperative seizures and reduce the amount of blood transfusions in patients who have cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Undergoing a cardiac surgical procedure (i.e., isolated CABG, isolated single cardiac valve surgery or a combination of both or isolated ascending aorta replacement) with the use of cardiopulmonary bypass
3. Provide written informed consent

Exclusion Criteria:

1. Allergy to tranexamic acid
2. Fulfill any of the following transfusion risk factors (A-F):

   A. Emergency surgery B. History of bleeding disorder C. Inherited thromboembolic or hemorrhagic disease D. Infective endocarditis (active) E. Pre-operative thrombocytopenia (<50,000 platelets per µL) F. Pre-operative hemoglobin <110 g/L
3. Estimated glomerular filtration rate <30 mL/min (CKD-EPI equation) or on dialysis
4. Pre-operative hemoglobin >170 g/L
5. Expected circulatory arrest
6. Pregnancy or breast feeding
7. Previous enrollment in DEPOSITION trial
8. Refusal of blood products (e.g., Jehovah's Witnesses)
9. Isolated Pericardiectomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Measure the level of plasma TxA at 5 time points | From baseline to on arrival in the intensive care unit, 3 hours after arrival, 6 hours after arrival, and the next morning.
  Measure the level of plasma TxA at 5 time points: pre-operative, on arrival in the intensive care unit, 3 hours after arrival, 6 hours after arrival, and the next morning.

SECONDARY OUTCOMES:
Measure the clot lysis time (i.e., fibrinolytic activity) at 5 time points | From baseline to on arrival in the intensive care unit, 3 hours after arrival, 6 hours after arrival, and the next morning.
  Measure the clot lysis time (i.e., fibrinolytic activity) at 5 time points: pre-operative baseline, on arrival in the intensive care unit, 3 hours after arrival, 6 hours after arrival, and the next morning.
Measure the plasmin generation (i.e., fibrinolytic activity) at 5 time points | From baseline to on arrival in the intensive care unit, 3 hours after arrival, 6 hours after arrival, and the next morning.
  Measure the plasmin generation (i.e., fibrinolytic activity) at 5 time points: pre-operative baseline, on arrival in the intensive care unit, 3 hours after arrival, 6 hours after arrival, and the next morning.

OTHER OUTCOMES:
Feasibility outcome (study-level): mean enrollment rate of the study | Start of enrollment (date of first patient) to end of enrollment (date of last patient).
  Determine whether the mean enrolment rate of the trial (total number of patients recruited / total recruitment period in weeks) is 2 patients per week or more.
Feasibility outcome (study-level): crossover rate of the study | Start of enrollment (date of first patient) to end of enrollment (date of last patient).
  Determine whether the percentage of crossovers between groups (total number of patients with crossover / total number of patients recruited * 100) is less than 5%.
Feasibility outcome (study-level): percentage of data completion of the study | Start of enrollment (date of first patient) to end of enrollment (date of last patient).
  Determine whether the percentage of data completion (total number of patients with complete outcome data / total number of patients enrolled * 100) is more than 95%.
Proportion of patients experiencing an in-hospital seizure | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  Appropriate descriptive statistics will be provided.
Proportion of patients requiring any blood product transfusion | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  Appropriate descriptive statistics will be provided.
Proportion of patients requiring re-operation for bleeding or cardiac tamponade | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  Appropriate descriptive statistics will be provided.
Proportion of patients requiring a red blood cell transfusion | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  Appropriate descriptive statistics will be provided.
Proportion of patients requiring pericardiocentesis | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  Appropriate descriptive statistics will be provided.
Duration of intensive care unit stay | Number of hours in ICU are being collected at the Post-Operative Visit. Hour collection will start upon arrival at ICU post surgery and stop at ICU exit, up to 10 days maximum.
  Appropriate descriptive statistics will be provided.
Proportion of patients experiencing the composite outcome of death, non-fatal myocardial infarction, or stroke | Start of surgery to hospital discharge or 10 days maximum (whichever occurs first)
  Appropriate descriptive statistics will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lamy, MD, Principal Investigator — Hamilton General Hospital
Locations (1):
- Hamilton Health Sciences - General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Habbab LM, Hussain S, Power P, Bashir S, Gao P, Semelhago L, VanHelder T, Parry D, Chu V, Lamy A. Decreasing Postoperative Blood Loss by Topical vs. Intravenous Tranexamic Acid in Open Cardiac Surgery (DEPOSITION) study: Results of a pilot study. J Card Surg. 2019 May;34(5):305-311. doi: 10.1111/jocs.14027. Epub 2019 Mar 25. PMID 30908754
- [Background] Lamy A, Sirota DA, Jacques F, Poostizadeh A, Noiseux N, Efremov S, Demers P, Akselrod B, Wang CY, Arora RC, Branny P, McGuinness SP, Brown CD, Jeanmart H, Zhao Q, Zhang H, Belley-Cote EP, Whitlock RP, Browne A, Copland I, Vincent J, Khatun R, Balasubramanian K, Bangdiwala SI, McGillion MH, Fox-Robichaud AE, Spence J, Yusuf S, Devereaux PJ; DEPOSITION Study Group. Topical Versus Intravenous Tranexamic Acid in Patients Undergoing Cardiac Surgery: The DEPOSITION Randomized Controlled Trial. Circulation. 2024 Oct 22;150(17):1315-1323. doi: 10.1161/CIRCULATIONAHA.124.069606. Epub 2024 Apr 8. PMID 38587333